CLINICAL TRIAL: NCT01498731
Title: The Effect of Integrating the Biomarker Copeptin Into the Process of Managing Patients With Suspected ACS
Brief Title: Effect of the Biomarker Copeptin in Managing Patients With Suspected Acute Coronary Syndrome (ACS)
Acronym: BiC-8
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Kerckhoff Klinik (Other); Heidelberg University (Other); Universitätsklinikum Hamburg-Eppendorf (Other); Wilhelminenspital Vienna (Other); University Hospital, Basel, Switzerland (Other)
Responsible Party: Principal Investigator, Martin Moeckel, Head Emergency Medicine, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Charite-BiC-8; DRKS00000276 (Other: German Clinical Trials Register); U1111-1118-1665 (Registry Identifier: International Clinical Trials Registry Platform)
Record Dates: First submitted 2011-10-25; First posted 2011-12-23 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-06

CONDITIONS: Acute Myocardial Infarction
Keywords: Copeptin; Troponin; Acute Coronary Syndrome; Rule-out of acute myocardial infarction; Emergency Medicine
MeSH Terms: conditions — Diabetes Insipidus; Acute Coronary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Copeptin (Experimental): Patients who test negative for Copeptin at admission will be considered low-risk and will be discharged home without further interventions.
  To secure the patients safety they will be transferred into our co-operating network of resident cardiologists using the software "Praxis-connect" i.e. these patients will be discharged with an electronically booked appointment to see a cardiologist preferably the next day (but latest within the next three days). In case of any findings suggestive of acute coronary syndrome or worsening of the patient's condition, the patient will immediately be re-admitted to our Emergency Room.
  Patients who test positive for Copeptin will be treated as by standard practise.
  Interventions: Behavioral: Discharge home
- Standard (No Intervention): Patients will be managed as by standard practice abiding current guidelines for the management of patients with suspected ACS.The copeptin result will not be available for the treating physician.

INTERVENTIONS:
Behavioral: Discharge home — Patients who test negative for Copeptin at admission will be considered low-risk and will be discharged home. To secure the patients safety they will be transferred into our co-operating network of resident cardiologists preferably the next day (but latest within the next three days). In case of any findings suggestive of acute coronary syndrome or worsening of the patient's condition, the patient will immediately be re-admitted to our Emergency Room.
  Arms: Copeptin

SUMMARY:
Acute chest pain is commonly known to be the classic symptom of acute myocardial infarction. Of the many patients which visit the Emergency Department because of chest pain, less than half do actually suffer from an acute myocardial infarction or acute myocardial ischemia. In some patients the acute myocardial infarction can be diagnosed at admission, either because of typical changes in their ECG (STEMI, ST-elevation myocardial infarction)or because of increased levels of the laboratory value Troponin in their blood (NSTEMI, Non-ST-elevation myocardial infarction). Troponin is currently the most important marker to diagnose acute myocardial infarction. Unfortunately a lot of patients with suspected acute coronary syndrome do not show any ECG or Troponin changes. These patients pose a major problem in emergency medicine as they need to precautionally be admitted to a chest pain unit and to be started on medical treatment until a second Troponin test after 6-9 hours is available.

In this study, we investigate the biomarker Copeptin. Copeptin has shown excellent results in diagnostic clinical trials assessing its use in various acute diseases. There are three important trials showing an excellent negative predictive value of Copeptin in combination with Troponin in patients with suspected acute coronary syndrome (Reichlin et al., JACC, 2009; Keller et al. JACC, 2010, Giannitsis et al. Clin Chem 2011).

This trial compares two processes of managing patients with suspected acute coronary syndrome (ACS), the standard process according to current guidelines and the experimental process integrating copeptin as a rule-out marker for acute myocardial infarction into management decisions. Main Hypothesis: Patients with suspected ACS who test negative for Troponin and negative for Copeptin at their initial presentation to the ED can safely be discharged (interventional process). They will not experience more major cardiac adverse events than patients who were managed by standard practise (control process)within 30 days after admission.

The Investigators want to test Copeptin in patients with suspected acute coronary syndrome in whom the ECG is unspecific and the initial Troponin test is negative. Further patient care will be based on the Copeptin result. Patients with a negative Copeptin will be discharged into the ambulant care of resident cardiologists.Copeptin positive patients will be managed according to standard guidelines for the management of patients with ACS.

DETAILED DESCRIPTION:
The management of patients with suspected Non-ST elevation acute coronary syndrome (NSTEACS) can be time-consuming and expensive. Often patients need to be hospitalized for precautionary medical treatment and serial Troponin testing until further decisions can be made.

Copeptin, a 39 amino acid glycopeptide, is the C-terminal portion of Pro-Vasopressin. It is co-secreted from the posterior pituitary gland together with Vasopressin and mirrors the amount of Vasopressin in the circulation. Vasopressin is primarily known as Anti-Diuretic Hormone (ADH), which acts in the kidney to regulate the body's retention of water and in high concentration causes arterial vasoconstriction.

Vasopressin is, as a central hormone, also a crucial part of the hypothalamo-pituitary-adrenal axis, which responds to severe, life-threatening "stress inputs"; its levels reflect the body's individual stress level.Vasopressin itself has a half-life of 5-10 minutes and is therefore difficult to measure in-vivo. Copeptin is secreted stoichiometrically with Vasopressin, it remains stable for days after blood withdrawal and can therefore easily be measured. Copeptin has been studied as a diagnostic and prognostic marker since 2006. In acute myocardial infarction Copeptin levels have been shown to increase early after the onset of symptoms (0-4 hours) and start decreasing after 4-5 hours.

In acute myocardial infarction (AMI) Copeptin levels increase early after the onset of symptoms. In patients with suspected ACS Copeptin levels were significantly higher in patients with AMI than in patients with other diagnoses. Copeptin in conjunction with Troponin T was particularly useful as a rule-out marker of AMI.

This is a randomized controlled diagnostic trial to quantify the benefit of integrating Copeptin into the management process of patients with NSTEACS and a negative baseline Troponin I test result in the Chest Pain Unit (CPU). Patient management will depend on Copeptin rather than serial Troponin results. Patients will be randomized in either a standard group (management according to current guidelines on managing patients with ACS, Copeptin will be tested, but result will not be revealed to treating personnel) or an interventional group (Copeptin testing, further management dependent on Copeptin result).

In this interventional group, patients with a negative baseline Copeptin will be discharged into the ambulant care of co-operating resident cardiologists. Patients with a positive Copeptin result will be treated as by standard care (like patients in the control group).

The investigators will assess the efficacy and safety of the new process as compared to the standard process. Secondary endpoints will assess patient satisfaction and length of hospital stay. This study design will not only assess the diagnostic use but also the clinical relevance of Copeptin testing in the ED/CPU.

Consecutive N-STEACS patients of the Chest Pain Unit with a negative Troponin I at admission will be invited to participate. Troponin I is tested as part of the standard management of patients with suspected acute coronary syndrome on a point of care test device (POCT).

Patients who give their written informed consent will then be randomized into one of two study arms (experimental and standard management) where further management depends on their Copeptin result at admission.

ELIGIBILITY:
Inclusion Criteria:

* Typical chest pain (with or without ECG-changes, but no ST-elevation)suggestive of unstable angina or non-ST-elevated myocardial infarction (NSTEMI)
* Troponin negative at admission according to the current clinical practice Patient willing and able to give written informed consent

Exclusion Criteria:

* Patients with ST-elevation myocardial infarction (STEMI)
* Continuing chest pain or recurrent episodes of chest pain under therapy
* High-risk patients with suspected ACS who need to be hospitalized for reasons independent of their initial troponin result
* Patients who need to be hospitalized for other medical reasons
* Patients in need of urgent life-saving interventions
* Patients under 18 years of age
* Patients with a life expectancy < 6 months
* Patients with any condition that leads the treating physician to not consider the patient eligible for the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 902 (Actual)
Dates: Start 2011-04; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Rate of major adverse cardiac events (MACE) within 30 days Copeptin vs. Control arm. | 30 days after discharge
  Rate of MACE (all- cause death or survived sudden cardiac arrest, myocardial infarction, re-hospitalisation for acute coronary syndrome, acute unplanned PCI, coronary artery bypass grafting (CABG) and documented life-threatening arrhythmias (VF, VT, AV-block III)) within 30 days Copeptin vs. Control arm (non-inferiority).

SECONDARY OUTCOMES:
Proportion of patients in whom coronary angiography (CA) is performed Copeptin vs. Control arm. | within 30 days after discharge
  Efficacy endpoint
  * Rate of Patients in whom CA is performed
  * Rate of Patients with PCI after Index CA
  * Rate of Patients with CABG after Index CA
Rate of ALL major adverse cardiac events (MACE) | 90 days after discharge
  Rate of ALL MACE at 90 days
  * all- cause death or survived sudden cardiac arrest
  * myocardial infarction
  * re-hospitalisation for acute coronary syndrome
  * acute unplanned PCI
  * coronary artery bypass grafting (CABG)
  * documented life-threatening arrhythmias (VF, VT, AV-block III)
Patient satisfaction regarding management within the ED/CPU | no specific time frame, before discharge
  Patient satisfaction regarding management before discharge from ED/CPU
Length of hospital stay | within 30 days after discharge
  Duration of hospital stay
  * Length of stay at the Emergency Room
  * Length of hospital stay in the CPU
  * Length of stay in an intensive care unit (ICU)
  * Total length of hospital stay in hours including time as an inpatient on other wards

CONTACTS AND LOCATIONS:
Overall Officials: Martin Möckel, MD, PhD, Principal Investigator — Charité - Universitätsmedizin Berlin, Berlin, Germany
Locations (6):
- Wilhelminenspital Vienna, Vienna, Austria
- Germany (4):
  - Kerckhoff-Klinik GmbH, Bad Nauheim
  - Charité - Universitätsmedizin Berlin, Berlin
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Universitätsklinikum Heidelberg, Heidelberg
- University Hospital Basel, Basel, Switzerland

REFERENCES:
- [Background] Mockel M, Muller R, Vollert J, Muller C, Danne O, Gareis R, Stork T, Dietz R, Koenig W. Lipoprotein-associated phospholipase A2 for early risk stratification in patients with suspected acute coronary syndrome: a multi-marker approach: the North Wuerttemberg and Berlin Infarction Study-II (NOBIS-II). Clin Res Cardiol. 2007 Sep;96(9):604-12. doi: 10.1007/s00392-007-0540-x. Epub 2007 Jun 27. PMID 17593313
- [Background] Thygesen K, Alpert JS, White HD; Joint ESC/ACCF/AHA/WHF Task Force for the Redefinition of Myocardial Infarction. Universal definition of myocardial infarction. Eur Heart J. 2007 Oct;28(20):2525-38. doi: 10.1093/eurheartj/ehm355. No abstract available. PMID 17951287
- [Background] Newby LK, Storrow AB, Gibler WB, Garvey JL, Tucker JF, Kaplan AL, Schreiber DH, Tuttle RH, McNulty SE, Ohman EM. Bedside multimarker testing for risk stratification in chest pain units: The chest pain evaluation by creatine kinase-MB, myoglobin, and troponin I (CHECKMATE) study. Circulation. 2001 Apr 10;103(14):1832-7. doi: 10.1161/01.cir.103.14.1832. PMID 11294799
- [Background] Pope JH, Aufderheide TP, Ruthazer R, Woolard RH, Feldman JA, Beshansky JR, Griffith JL, Selker HP. Missed diagnoses of acute cardiac ischemia in the emergency department. N Engl J Med. 2000 Apr 20;342(16):1163-70. doi: 10.1056/NEJM200004203421603. PMID 10770981
- [Background] Itoi K, Jiang YQ, Iwasaki Y, Watson SJ. Regulatory mechanisms of corticotropin-releasing hormone and vasopressin gene expression in the hypothalamus. J Neuroendocrinol. 2004 Apr;16(4):348-55. doi: 10.1111/j.0953-8194.2004.01172.x. PMID 15089973
- [Background] Katan M, Morgenthaler N, Widmer I, Puder JJ, Konig C, Muller B, Christ-Crain M. Copeptin, a stable peptide derived from the vasopressin precursor, correlates with the individual stress level. Neuro Endocrinol Lett. 2008 Jun;29(3):341-6. PMID 18580851
- [Background] Khan SQ, Dhillon OS, O'Brien RJ, Struck J, Quinn PA, Morgenthaler NG, Squire IB, Davies JE, Bergmann A, Ng LL. C-terminal provasopressin (copeptin) as a novel and prognostic marker in acute myocardial infarction: Leicester Acute Myocardial Infarction Peptide (LAMP) study. Circulation. 2007 Apr 24;115(16):2103-10. doi: 10.1161/CIRCULATIONAHA.106.685503. Epub 2007 Apr 9. PMID 17420344
- [Background] Reichlin T, Hochholzer W, Stelzig C, Laule K, Freidank H, Morgenthaler NG, Bergmann A, Potocki M, Noveanu M, Breidthardt T, Christ A, Boldanova T, Merki R, Schaub N, Bingisser R, Christ M, Mueller C. Incremental value of copeptin for rapid rule out of acute myocardial infarction. J Am Coll Cardiol. 2009 Jun 30;54(1):60-8. doi: 10.1016/j.jacc.2009.01.076. PMID 19555842
- [Background] Voors AA, von Haehling S, Anker SD, Hillege HL, Struck J, Hartmann O, Bergmann A, Squire I, van Veldhuisen DJ, Dickstein K; OPTIMAAL Investigators. C-terminal provasopressin (copeptin) is a strong prognostic marker in patients with heart failure after an acute myocardial infarction: results from the OPTIMAAL study. Eur Heart J. 2009 May;30(10):1187-94. doi: 10.1093/eurheartj/ehp098. Epub 2009 Apr 3. PMID 19346228
- [Background] Keller T, Tzikas S, Zeller T, Czyz E, Lillpopp L, Ojeda FM, Roth A, Bickel C, Baldus S, Sinning CR, Wild PS, Lubos E, Peetz D, Kunde J, Hartmann O, Bergmann A, Post F, Lackner KJ, Genth-Zotz S, Nicaud V, Tiret L, Munzel TF, Blankenberg S. Copeptin improves early diagnosis of acute myocardial infarction. J Am Coll Cardiol. 2010 May 11;55(19):2096-106. doi: 10.1016/j.jacc.2010.01.029. PMID 20447532
- [Background] Morgenthaler NG, Struck J, Alonso C, Bergmann A. Assay for the measurement of copeptin, a stable peptide derived from the precursor of vasopressin. Clin Chem. 2006 Jan;52(1):112-9. doi: 10.1373/clinchem.2005.060038. Epub 2005 Nov 3. PMID 16269513
- [Background] Giannitsis E, Kehayova T, Vafaie M, Katus HA. Combined testing of high-sensitivity troponin T and copeptin on presentation at prespecified cutoffs improves rapid rule-out of non-ST-segment elevation myocardial infarction. Clin Chem. 2011 Oct;57(10):1452-5. doi: 10.1373/clinchem.2010.161265. Epub 2011 Aug 1. PMID 21807867
- [Derived] Giannitsis E, Garfias-Veitl T, Slagman A, Searle J, Muller C, Blankenberg S, von Haehling S, Katus HA, Hamm CW, Huber K, Vollert JO, Mockel M. Biomarkers-in-Cardiology 8 RE-VISITED-Consistent Safety of Early Discharge with a Dual Marker Strategy Combining a Normal hs-cTnT with a Normal Copeptin in Low-to-Intermediate Risk Patients with Suspected Acute Coronary Syndrome-A Secondary Analysis of the Randomized Biomarkers-in-Cardiology 8 Trial. Cells. 2022 Jan 8;11(2):211. doi: 10.3390/cells11020211. PMID 35053326
- [Derived] Reinhold T, Giannitsis E, Mockel M, Frankenstein L, Vafaie M, Vollert JO, Slagman A. Cost analysis of early discharge using combined copeptin/cardiac troponin testing versus serial cardiac troponin testing in patients with suspected acute coronary syndrome. PLoS One. 2018 Aug 23;13(8):e0202133. doi: 10.1371/journal.pone.0202133. eCollection 2018. PMID 30138394